CLINICAL TRIAL: NCT02536144
Title: The Clinical Application of Magnetic-controlled Capsule Endoscopy System in Examination of Human Colon
Brief Title: The Clinical Application of MCCES in Examination of Human Colon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: NFEK-2015-046
Record Dates: First submitted 2015-08-24; First posted 2015-08-31 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Abdominal Pain; Diarrhea; Hematochezia
Keywords: colon capsule; magnetic; maneuverability; colonoscopy
MeSH Terms: conditions — Abdominal Pain; Diarrhea; Gastrointestinal Hemorrhage | interventions — Colonoscopy; Colonoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCCES (Experimental): Magnetic -controlled capsule endoscopy system (MCCES) is a robot system that the capsule would be swallowed to observe the mucosa of the human alimentary canal especially the colon under the control of the magnetic-manipulator.
  Interventions: Procedure: magnetic-controlled capsule endoscopy system
- Colonoscopy (Active Comparator): Colonoscopy has now been in use for many years to visualize and diagnose abnormalities of the colon and it is the gold standard for detecting colorectal lesions.In this study,the additional utility of the colonoscopy is to monitor the movement of the Magnetic -controlled capsule endoscopy.
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: magnetic-controlled capsule endoscopy system — 1. A magnetic-controlled capsule endoscopy(MCCE) included camera,magnet,batter and high polymer material shell.
  2. The MCCE would be turned to sleeping mode capturing picture at a rate of 0.5 frame per second after being swallowed.
  3. While reaching cecum, the MCCE would be turned to a working mode capturing picture at a rate of 2 frame per second.
  4. The MCCE would be controlled by the Magnetic-manipulator out of body to finish the motion of e rotation, somersault, Bird's-eye view, worm's eye view from cecum to anus.
  Arms: MCCES
Procedure: Colonoscopy — 1. Bowel preparation should be well done before the examination.
  2. A tube with illumination and camera system would insert into colon from anus.
  3. From the pictures captured by the camera ,the doctor would see the mucous of the colon.
  Other Names: colonoscope
  Arms: Colonoscopy

SUMMARY:
This study is to determine the feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human colon under the real time monitoring by colonoscopy in the clinical application.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of cancer-related deaths in the Western world. The screening tests include flexible sigmoidoscopy, optical colonoscopy (OC), double-contrast barium enema , or CT colonography . Such screening can reduce CRC incidence and mortality but its effectiveness depends on its quality, ease of use, and patient adherence .Colon capsule endoscopy(CCE) is being actively evaluated as an emerging complementary or alternative procedure for evaluation of the colon. magnetic -controlled capsule endoscopy system is a new ingestible colon capsule robot provided by Chongqing Jinshan Science & Technology. While Screening the colon, the capsule is drove by magnetic-manipulator outside the body, which means it can move from the cecum to anus step by step under the control of the doctor. However, there's little data report on this colon capsule robot system in clinical application. The investigators plan to conduct this prospective study to determine the feasibility and safety of magnetic-controlled capsule endoscopy system in examination of human colon under the real time monitoring by colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients who repeatedly have the symptom such as abdominal pain, diarrhea, hematochezia and so on, or
* Patients who volunteer to the colonoscopy screening.

Exclusion Criteria:

* Dysphagia or swallowing disorder,
* Congestive heart failure,
* Renal insufficiency,
* Prior major abdominal surgery of the gastrointestinal tract,
* Known or suspected bowel obstruction,
* Presence of a cardiac pacemaker or other implanted electromedical devices,
* Allergy or contraindication to the medications used in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Maneuverability | From the MCCES examination began until the capsule excreted, an expected average of 24h
  The Maneuverability was defined as the rotation, somersault, Bird's-eye view, worm's eye view of the capsule, and completing any motion would gain 1 point, eventually ,4 point was good,2-3 point moderate,0-1point poor.

SECONDARY OUTCOMES:
Migration length of anus direction | From the MCCES examination began until the capsule excreted, an expected average of 24h
  Migration length of anus direction was defined as how long was the distance the capsule controlled by the Magnetic-manipulator moved from cecum to anus in 25 minutes.
The movement of mouth direction | From the MCCES examination began until the capsule excreted, an expected average of 24h
  The movement of mouth direction was defined as if the capsule controlled by the Magnetic-manipulator could move from any point of the colon towards mouth direction.
Nidus of colon | During the procedure
  From date of the examination until the date of pathological diagnosis, an expected average of 7 days
The level of cleanliness | From the MCCES examination began until the capsule excreted, an expected average of 24h
  The cleanliness of the colon was graded as excellent (No more than small bits of adherent feces),good(Small amount of feces or dark fluid,but not enough to interfere with the examination ),fair(Enough feces or dark fluid present to preclude a completely reliable examination),poor(large amount of fecal residue).
Procedure related complication | From the day of the examination until the follow up ended ,access up to 7 days.
  Perforation, capsule retention, abdominal pain and so .etc.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Jiang, doctor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Result] Spada C, Hassan C, Ingrosso M, Repici A, Riccioni ME, Pennazio M, Pirozzi GA, Pagano N, Cesaro P, Spera G, Petruzziello L, Costamagna G. A new regimen of bowel preparation for PillCam colon capsule endoscopy: a pilot study. Dig Liver Dis. 2011 Apr;43(4):300-4. doi: 10.1016/j.dld.2010.10.005. Epub 2010 Nov 18. PMID 21087902
- [Result] Hagel AF, Gabele E, Raithel M, Hagel WH, Albrecht H, de Rossi TM, Singer C, Schneider T, Neurath MF, Farnbacher MJ. Colon capsule endoscopy: detection of colonic polyps compared with conventional colonoscopy and visualization of extracolonic pathologies. Can J Gastroenterol Hepatol. 2014 Feb;28(2):77-82. doi: 10.1155/2014/691785. PMID 24501724
- [Derived] Gu H, Zheng H, Cui X, Huang Y, Jiang B. Maneuverability and safety of a magnetic-controlled capsule endoscopy system to examine the human colon under real-time monitoring by colonoscopy: a pilot study (with video). Gastrointest Endosc. 2017 Feb;85(2):438-443. doi: 10.1016/j.gie.2016.07.053. Epub 2016 Jul 29. PMID 27480288
- See also: Homepage of Department of Gastroenterology, Nanfang Hospital of Southern Medical University — http://www.nfyy.com/